CLINICAL TRIAL: NCT06245408
Title: A Phase 3 Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Dazodalibep in Participants With Sjögren's Syndrome With Moderate-to-Severe Symptom State (HZNP-DAZ-303)
Brief Title: A Safety and Efficacy Study of Dazodalibep in Participants With Sjögren's Syndrome (SS) With Moderate-to-Severe Symptom State
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HZNP-DAZ-303
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Sjögren's Syndrome (SS)
Keywords: European Alliance of Associations for Rheumatology Sjögren's Syndrome Disease Activity Index (ESSDAI); European Alliance of Associations for Rheumatology Sjögren's Syndrome Patient Reported Index (ESSPRI); European Alliance of Associations for Rheumatology (EULAR)
MeSH Terms: conditions — Sjogren's Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dazodalibep Dose 1 (Experimental): Participants will be administered dose 1 of dazodalibep by intravenous (IV) infusion.
  Interventions: Drug: Dazodalibep
- Dazodalibep Dose 2 (Experimental): Participants will be administered dose 2 of dazodalibep by IV infusion.
  Interventions: Drug: Dazodalibep
- Placebo (Placebo Comparator): Participants will be administered placebo by IV infusion.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dazodalibep — IV infusion
  Other Names: VIB 4920; MEDI4920
  Arms: Dazodalibep Dose 1; Dazodalibep Dose 2
Drug: Placebo — IV infusion
  Arms: Placebo

SUMMARY:
Primary Objective:

To evaluate the effect of dazodalibep on patient-reported symptoms of SS in participants with moderate-to-severe symptom state

Secondary Objectives:

1. To evaluate the effect of dazodalibep on patient-reported outcomes (PROs) in participants with SS.
2. To evaluate the effect of dazodalibep on measures of systemic activity, PROs, and salivary flow in participants with SS
3. To evaluate the safety and tolerability of multiple doses of dazodalibep in participants with SS

DETAILED DESCRIPTION:
Acquired from Horizon in 2024.

ELIGIBILITY:
Key Inclusion Criteria:

1. Diagnosed with SS by meeting the 2016 ACR/EULAR Classification Criteria
2. Have an ESSPRI score of ≥ 5 at screening.
3. Have an ESSDAI score of < 5 at screening.
4. Positive for either anti-Ro autoantibodies or RF, or both at screening (as per the definition of the standard central laboratory test).
5. Residual salivary gland function as defined by whole stimulated salivary flow > 0.1 mL/min.
6. Vaccinated against SARS-CoV-2 according to current local authority guidelines at least 2 weeks prior to screening unless participant refuses vaccination.
7. Meets all of the following tuberculosis (TB) criteria:

   1. No history of latent or active TB prior to screening, except for latent TB with documented completion of locally appropriate treatment.
   2. No signs or symptoms suggestive of active TB from medical history or physical examination.
   3. No recent (≤ 12 weeks of screening) close contact with a person with active TB (close contact is defined as ≥ 4 hours/week OR living in the same household OR in a house where a person with active TB is a frequent visitor).
   4. Negative Interferon Gamma Release Assay (IGRA) test result for TB at screen unless previously treated as per Inclusion Criterion. Participants with an indeterminate test result can repeat the test, but if the repeat test is also indeterminate, they are excluded.
   5. A chest radiograph (obtained during the screening period or any time within 12 weeks prior to screening) with no evidence of current active TB or other infection, or prior TB, malignancy, or clinically significant abnormalities suggesting an active process (unless due to SS).

Key Exclusion Criteria:

1. Individuals with medical history of confirmed deep venous thrombosis, pulmonary embolism, or arterial thromboembolism within 2 years of screening.
2. History or presence of concomitant polymyositis or dermatomyositis or systemic sclerosis.
3. Active malignancy or history of malignancy within the last 5 years, except as follows:

   1. In situ carcinoma of the cervix treated with apparent success with curative therapy > 12 months prior to screening; OR
   2. Cutaneous basal cell carcinoma following presumed curative therapy.
4. Individuals who are pregnant or lactating or planning to become pregnant during the study.
5. Individuals with known history of severe allergy or reaction to any component of the IP formulation or to any other biologic therapy.
6. Individuals with any severe cardiovascular, respiratory, endocrine, gastrointestinal, hematological, neurological, psychiatric, or systemic disorder or any other condition that, in the opinion of the Investigator, would place the individual at unacceptable risk of complications, interfere with evaluation of the IP, or confound the interpretation of participant safety or study results.
7. Individuals who have a positive test for, or have been treated for, hepatitis B, hepatitis c or HIV infection.
8. Individuals with a positive test for SARS-CoV-2 on the day of randomization or symptoms suggestive of SARS-CoV-2 at randomization or significant exposure to coronavirus disease 2019 (COVID-19) within 10 calendar days prior to randomization.
9. Individuals with:

   1. A history of more than one episode of herpes zoster and/or opportunistic infections in the last 12 months, with the exception of non-invasive herpes simplex at any site, oral candidiasis, vaginal candidiasis, or cutaneous fungal infections, which are permitted within the prior 12 months unless of unusual severity.
   2. Active infection requiring systemic treatment at the time of screening or through randomization, or history of more than 2 infections requiring IV antibiotics within 12 months prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 434 (Actual)
Dates: Start 2024-04-08 (Actual); Primary Completion 2026-10-22 (Estimated); Study Completion 2026-12-17 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in ESSPRI score | At Week 48
Change from baseline in Diary for Assessing Sjogren's Patient Reported Index (DASPRI ) score | At week 48

SECONDARY OUTCOMES:
Proportion of participants achieving meaningful improvement in DASPRI | At Week 48
Proportion of participants achieving ESSPRI [1.5] response | At Week 48
Change from baseline in Patient-Reported Outcomes Measurement Information System Fatigue-Short Form 10a (PROMIS-Fatigue SF-10a) | At Week 48
Change from baseline in DASPRI Dryness | At Week 48
Change from baseline in ESSPRI Dryness | At Week 48
Change from baseline in DASPRI Pain | At Week 48
Change from baseline in ESSPRI Pain | At Week 48
Change from baseline in 36-item Short Form Survey (SF-36) Physical Component Summary (PCS) score | At Week 48
Change from baseline in DASPRI total score | At week 12 and week 24
Change from baseline in ESSPRI total score | At week 12, Week 24
Change from baseline in DASPRI Fatigue | At Week 48
Change from baseline in ESSPRI fatigue domain score | At Week 48
Change from baseline in total stimulated salivary flow | At Week 48
Number of participants With Treatment Emergent Adverse Events (TEAEs) | Baseline (Day 1) to Week 56
Number of participants With Treatment Emergent Serious Adverse Events (TESAEs) | Baseline (Day 1) to Week 56
Number of participants With Adverse Events of Special Interest (AESIs) | Baseline (Day 1) to Week 56

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (194):
- United States (41):
  - Arizona Arthritis & Rheumatology Associates - Avondale, Avondale, Arizona
  - Arizona Research Clinic PLLC, Chandler, Arizona
  - Arizona Arthritis and Rheumatology Associates - Flagstaff - 399 S Malpais Ln, Flagstaff, Arizona
  - Arizona Arthritis and Rheumatology Associates - Gilbert - 3645 S Rome St, Gilbert, Arizona
  - Arizona Arthritis and Rheumatology Associates - Glendale - 5681 W Beverly Ln, Glendale, Arizona
  - Arizona Arthritis and Rheumatology Associates - Tucson - 2001 W Orange Grove Rd, Tucson, Arizona
  - Medvin Clinical Research - Covina, Covina, California
  - UCSD Altman Clinical and Translational Research Institute Building, La Jolla, California
  - Inland Rheumatology Clinical Trials Incorporated, Upland, California
  - Medvin Clinical Research, Whittier, California
  - Tekton Research, LLC - 2121 E Harmony Rd - PPDS, Fort Collins, Colorado
  - Bradenton Research Center Inc, Bradenton, Florida
  - Clinical Research of West Florida Inc - Clearwater, Clearwater, Florida
  - West Broward Rheumatology Associates, Inc., Tamarac, Florida
  - BayCare Medical Group Primary Care and Rheumatology - Tampa, Tampa, Florida
  - University of Kansas Medical Center, Kansas City, Kansas
  - Tufts Medical Center - Rheumatology Research Office - PPDS, Boston, Massachusetts
  - Clinical Research Institute of Michigan, LLC-St. Claire Shores, Saint Clair Shores, Michigan
  - Kansas City Physician Partners-8350 N Saint Clair Ave, Kansas City, Missouri
  - Arthritis, Rheumatic & Bone Disease Associates - P, Voorhees Township, New Jersey
  - Albuquerque Center for Rheumatology, Albuquerque, New Mexico
  - NYU Langone Health - Joseph S. and Diane H. Steinberg Ambulatory Care Center, Brooklyn, New York
  - Arthritis and Osteoporosis Consultants of The Carolinas, Charlotte, North Carolina
  - Duke Early Phase Clinical Research Unit - PPDS, Durham, North Carolina
  - Onsite Clinical Solutions, LLC - Salisbury, Salisbury, North Carolina
  - Arthritis & Osteoporosis Center of Southwest Ohio - Miamisburg, Miamisburg, Ohio
  - University of Toledo Medical Center, Toledo, Ohio
  - STAT Research-600 Aviator Ct, Vandalia, Ohio
  - Low Country Rheumatology PA-Summerville, Summerville, South Carolina
  - Murfreesboro Medical Clinic Westlawn, Murfreesboro, Tennessee
  - Amarillo Center For Clinical Research, Amarillo, Texas
  - Accurate Clinical Management-Baytown, Baytown, Texas
  - Precision Comprehensive Clinical Research Solutions, Grapevine, Texas
  - R & H Clinical Research-777 S Fry Rd, Katy, Texas
  - Texas Arthritis & Rheumatology Associates, Katy, Texas
  - Valley Arthritis Center, McAllen, Texas
  - University of Texas - San Antonio - Health Science Center - PPDS, San Antonio, Texas
  - Advanced Rheumatology of Houston - The Woodlands, The Woodlands, Texas
  - DM Clinical Research - Migraine and COPD - PPDS, Tomball, Texas
  - Western Washington Medical Group, Bothell, Washington
  - Rheumatology and Pulmonary Clinic, Beckley, West Virginia
- Argentina (15):
  - Sanatorio Agote - Swiss Medical Group - PPDS, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Sanatorio Guemes, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Framingham Centro Médico, La Plata, Buenos Aires
  - Instituto CER S.A., Quilmes, Buenos Aires
  - Instituto de Investigaciones Clinicas Quilmes SRL, Quilmes, Buenos Aires
  - Hospital General de Agudos Dr. José María Ramos Mejia, Buenos Aires, Ciudad Autónoma de BuenosAires
  - Consultorios Médicos Dr. Doreski - Fundacion Respirar - PPDS, Buenos Aires, Ciudad Autónoma de BuenosAires
  - Centro de Investigaciones Médicas Tucumán - PPDS, San Miguel de Tucumán, Tucumán Province
  - Centro de Investigaciones Reumatológicas, San Miguel de Tucumán, Tucumán Province
  - Clínica Mayo de U.M.C.B. S.R.L, San Miguel de Tucumán, Tucumán Province
  - DOM Centro de Reumatología, Buenos Aires
  - Aprillus Asistencia e Investigacion de Arcis Salud SRL, Buenos Aires
  - Centro Medico Arsema, Buenos Aires
  - Sanatorio Allende S.A, Córdoba
  - Centro Polivalente de Asistencia e Investigación Clínica - CER San Juan, San Juan
- The Queen Elizabeth Hospital, Woodville South, South Australia, Australia
- UZ Gent, Ghent, Belgium
- Brazil (4):
  - SER - Serviços Especializados em Reumatologia da Bahia S/S - ME, Salvador, Estado de Bahia
  - Irmandade da Santa Casa de Misericórdia de Belo Horizonte - PPDS, Belo Horizonte, Minas Gerais
  - Centro de Estudos em Terapias Inovadoras, Curitiba, Paraná
  - LMK Servicos Medicos SS, Porto Alegre, Rio Grande do Sul
- Centre de Recherche Musculo-Squelettique - 1920 Rue Bellefeuille, Trois-Rivières, Quebec, Canada
- Chile (4):
  - Clinical Research Chile SpA - PPDS, Valdivia, Los Ríos Region
  - Centro de Investigacion de Enfermedades Respiratorias e inmunologicas, Viña del Mar, Región de Valparaíso
  - BIOCINETIC Ltda, Peñalolén, Región-MetropolitanadeSantiago
  - Enroll SpA - Dr. Manuel Barros Borgono - PPDS, Santiago, Región-MetropolitanadeSantiago
- Croatia (5):
  - Clinical Center Zagreb - Oncology - Salata 7 - PPDS, Zagreb, City of Zagreb
  - Clinical Hospital Sveti Duh, Zagreb, City of Zagreb
  - Polyclinic Bonifarm, Zagreb, City of Zagreb
  - Clinical Hospital Centre Osijek, Osijek
  - University Hospital of Split-Spinciceva 1, Split
- France (5):
  - CHU de Bordeaux - Hôpital Saint-André, Bordeaux
  - CHU de Brest - Hôpital La Cavale Blanche, Brest
  - Hopital Emile Muller, Mulhouse
  - AP-HP - Hôpital Saint Antoine, Paris
  - Hôpitaux Universitaires de Strasbourg, Strasbourg
- Germany (5):
  - University Clinic Heidelberg, Heidelberg, Baden-Wurttemberg
  - Rheumazentrum Prof. Dr. med. Gunther Neeck-Standort Bad Doberan, Bad Doberan, Mecklenburg-Vorpommern
  - Rheumazentrum Greifswald, Greifswald Hansestadt, Mecklenburg-Vorpommern
  - DRK Gemeinnützige Krankenhaus GmbH Sachsen - DRK Krankenhaus Chemnitz-Rabenstein, Chemnitz
  - MVZ Rheuma, Hamburg
- Greece (3):
  - Laiko General Hospital of Athens, Athens, Attica
  - University General Hospital of Larissa, Larissa, Larisa
  - Euromedica Kianous Stavros, Thessaloniki
- Hungary (3):
  - Bekes Varmegyei Kozponti Korhaz, Gyula, Bekes County
  - Vasarhelyi Sarkanyfu Kft., Hódmezővásárhely, Csongrád megye
  - Del-pesti Centrumkorhaz- Orszagos Hematologiai és Infektologiai Intezet - Albert Flórián út 5-7, Budapest
- Italy (10):
  - AUSL di Reggio Emilia - IRCCS - Arcispedale Santa Maria Nuova, Reggio Emilia, Emilia-Romagna
  - Azienda Sanitaria Universitaria Friuli Centrale - PO Universitario Santa Maria della Misericordia, Udine, Friuli Venezia Giulia
  - Fondazione Policlinico Universitario Campus Bio-Medico, Rome, Lazio
  - Fondazione Policlinico Universitario A Gemelli - Rome - PPDS, Rome, Lazio
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan, Lombardy
  - Azienda Ospedaliero Universitaria Maggiore della Carità, Novara, Piedmont
  - Azienda Ospedaliera Universitaria Careggi, Florence, Tuscany
  - Azienda Ospedaliera Universitaria Integrata Di Verona, Verona, Veneto
  - AOU Policlinico Gaspare Rodolico-San Marco - Presidio Ospedaliero San Marco, Catania
  - Azienda Ospedaliero Universitaria Pisana - Stabilimento Santa Chiara, Pisa
- Japan (22):
  - Chubu Rosai Hospital, Nagoya, Aiti
  - Japan Community Health Care Organization (JCHO) Chukyo Hospital, Nagoya, Aiti
  - Daido Clinic, Nagoya, Aiti
  - Sapporo Medical University Hospital, Sapporo, Hokkaidô
  - Hokkaido University Hospital, Sapporo, Hokkaidô
  - Hospital of the University of Occupational and Environmental Health, Japan, Kita Kyushu-shi, Hukuoka
  - Hyogo Medical University Hospital, Nishinomiya-Shi, Hyôgo
  - University of Tsukuba Hospital, Tsukuba, Ibaraki
  - Kanazawa Medical University Hospital, Kahoku, Ishikawa-ken
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - National Hospital Organization Yokohama Medical Center, Yokohama, Kanagawa
  - University Hospital, Kyoto Prefectural University of Medicine, Kyoto, Kyôto
  - Kyoto University Hospital, Kyoto, Kyôto
  - Nagasaki University Hospital, Nagasaki, Nagasaki
  - Sasebo Chuo Hospital, Sasebo-Shi, Nagasaki
  - Kurashiki Medical Clinic, Kurashiki-Shi, Okayama-ken
  - Saitama Medical University Hospital, Iruma-gun, Saitama
  - Hamamatsu University Hospital, Hamamatsu, Shizuoka
  - St. Luke's International Hospital, Chuo-Ku, Tokyo
  - Tokyo Medical Center, Meguro-Ku, Tokyo
  - Keio University Hospital, Shinjuku-Ku, Tokyo
  - Nihon University Itabashi Hospital, tabashi City, Tokyo
- Mexico (11):
  - Mediadvance Clinical S.A.P.I. de C.V., Parques de San Felipe, Chihuahua
  - CIMAB SA de CV, Torreón Centro, Coahuila
  - Centro de Investigación en Artritis y Osteoporosis - PPDS, Mexicali, Estado de Baja California
  - Bioclinica - Centro Integral En Reumatologia Sociedad Anónima de Capital Variable - PPDS, Americana, Jalisco
  - Cryptex Investigación Clínica, S.A. de C.V., Mexico City, Mexico City
  - Centro de Investigación y Tratamiento Reumatológico S.C, San Miguel Chapultepec, Mexico City
  - Oaxaca Site Management Organization - Clinic - OSMO - PPDS, Centro, Oaxaca
  - Consultorio de Reumatologia, México
  - Clinstile, S.A. de C.V., México
  - Hospital Universitario Dr. Jose Eleuterio González, Mitras Centro
  - Accelerium, S. de R.L. de C.V. - PPDS, Monterrey
- New Zealand (3):
  - Optimal Clinical Trials Ltd - PPDS, Auckland, North Island
  - Aotearoa Clinical Trials Trust, Auckland
  - Waikato Hospital, Hamilton
- Peru (8):
  - Clinica San Antonio S.A.C, Trujillo, La Libertad
  - Clinica San Juan Bautista, San Juan de Lurigancho, Lima region
  - Hogar Clinica San Juan de Dios - Arequipa, Arequipa
  - Hospital Militar Central Luis Arias Schereiber, Lima
  - Clínica Internacional San Borja-Avenida Guardia Civil 385, Lima
  - Instituto Peruano del Hueso y la Articulacion S.A.C., Lima
  - Instituto de Ginecologia y Reproduccion - PPDS, Lima
  - Alfredo Berrocal Kasay Reuma Sociedad de Responsabilidad Limitada, Pueblo Libre
- Poland (20):
  - Malopolskie Centrum Kliniczne, Krakow, Lesser Poland Voivodeship
  - FutureMeds - Wroclaw - PPDS, Wroclaw, Lower Silesian Voivodeship
  - Centrum Medyczne Oporow, Wroclaw, Lower Silesian Voivodeship
  - ETG Lublin - PPDS, Lublin, Lublin Voivodeship
  - Reumed Sp. z o.o., Lublin, Lublin Voivodeship
  - FutureMeds - Warszawa Centrum - PPDS, Warsaw, Masovian Voivodeship
  - MICS Centrum Medyczne Warszawa - MICS - PPDS, Warsaw, Masovian Voivodeship
  - MTZ Clinical Research Powered by PRATIA - PPDS, Warsaw, Masovian Voivodeship
  - Narodowy Instytut Geriatrii, Reumatologii i Rehabilitacji im. Prof. Dr hab. Med. Eleonory Reicher, Warsaw, Masovian Voivodeship
  - Klinika Reuma Park sp . zoo Sp.k., Warsaw, Masovian Voivodeship
  - K2J2 Medical Center, Wołomin, Masovian Voivodeship
  - Centrum Badawcze Panaceum Agnieszka Brzezicka Magdalena Lenkiewicz Sp. Z o.o., Malbork, Pomeranian Voivodeship
  - Szpital Uniwersytecki Nr 2 im. Dr Jana Biziela w Bydgoszczy, Bydgoszcz
  - Centrum Medyczne Pratia Katowice - PPDS, Katowice
  - Centrum Medyczne Plejady Magdalena Celinska - Lowenhoff, Michal Zolnowski Spolka komandytowa, Krakow
  - FutureMeds - Lodz - PPDS, Lodz
  - Twoja Przychodnia PCM, Poznan
  - WIM-PIB, Centralny Szpital Kliniczny MON, Warsaw
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza Radeckiego we Wroclawiu - Borowska 213, Wroclaw
  - Pracownia Badan Klinicznych Salus - ul. Ołtaszyńska 92c/3, Wroclaw
- Portugal (4):
  - ULS de Lisboa Ocidental, EPE - Hospital Egas Moniz, Lisbon
  - Centro Hospitalar Universitário Lisboa Norte, E.P.E - PPDS, Lisbon
  - Hospital Conde de Bertiandos - Unidade Local de saúde do Alto Minho, EPE - Ponte de Lima, Ponte de Lima
  - ULS de Gaia/Espinho, EPE - Unidade I, Vila Nova de Gaia
- GCM Medical Group, PSC -62 Calle Jose Marti, San Juan, Puerto Rico
- Serbia (6):
  - Institute of Rheumatology - PPDS, Belgrade
  - Military Medical Academy, Belgrade
  - University Clinical Center of Serbia - Pasterova 2 - PPDS, Belgrade
  - University Clinical Center Kragujevac, Kragujevac
  - Clinical Centre of Vojvodina, Novi Sad
  - Special Hospital For Rheumatic Diseases Novi Sad, Novi Sad
- Slovenia (2):
  - University Medical Centre Ljubljana-Vodnikova cesta 62, Ljubljana
  - University Clinical Centre Maribor, Maribor
- South Korea (2):
  - Chonnam National University Hospital, Gwangju
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
- Spain (11):
  - C.H. Regional Reina Sofia - PPDS, Córdoba, Córdoba
  - Hospital Universitario de Basurto, Bilbao, Vizcaya
  - Hospital Universitario A Coruña, A Coruña
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz - PPDS, Madrid
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna
  - Fundacio Hospital de l'Esperit Sant, Santa Coloma de Gramenet(Barcelona)
  - Hospital Quironsalud Infanta Luisa, Seville
  - Hospital Nuestra Señora de Valme, Seville
  - Hospital Universitario Araba - Txagorritxu, Vitoria-Gasteiz, Álava
- Taiwan (4):
  - Kaohsiung Medical University - Chung-Ho Memorial Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - Taipei Medical University Hospital - PPDS, Taipei
  - Chang Gung Memorial Hospital, Linkou, Taoyuan
- United Kingdom (2):
  - Chapel Allerton Hospital - PPDS, Leeds
  - William Harvey Research Institute - PPDS, London

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com